CLINICAL TRIAL: NCT03974477
Title: Randomized Controlled Trial With SALT CONTROL H - Impact on Individual Sodium and Sodium to Potassium Ratio Excretion
Brief Title: Study With an Innovative Equipment to Monitor and Control SALT During Cooking
Acronym: iMC_SALT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: Fundação para a Ciência e a Tecnologia (Other); Instituto Nacional de Saúde Doutor Ricardo Jorge (Unknown); Centro Hospitalar De São João, E.P.E. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: iMCSALT19-21
Record Dates: First submitted 2019-04-29; First posted 2019-06-05 (Actual); Last update posted 2021-01-08 (Actual); Status verified 2020-12

CONDITIONS: Salt; Excess; Hypertension
Keywords: Dietary Salt; Urinary sodium excretion; Cooking; Hypertension; Randomized Controlled Trial; Sodium; Diet; Patient Education
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention will last for 8 weeks, an individual session of presentation of SALT CONTROL H will be carried out, with explanation of how the equipment works in the culinary preparation with an adequate salt content (will be used an illustrative video and recipes with an adequate salt content); use of SALT CONTROL H at home by the participant to control the use of salt during the cooking process; supervision and enhancement of the use of equipment; daily occurrence log; and the application of a satisfaction questionnaire on the use of SALT CONTROL H. A leaflet will also be delivered about "The new Food Wheel, a guide to the daily food choice!".
  Interventions: Device: SALT CONTROL H equipment to control and monitor salt during cooking process
- Control (No Intervention): No intervention will be carried out except the provision of a leaflet on "The new Food Wheel, a guide to the daily food choice!" to the participants.

INTERVENTIONS:
Device: SALT CONTROL H equipment to control and monitor salt during cooking process — Participants will use SALT CONTROL H at home during 8 weeks to cook meals with adequate salt content.
  Arms: Intervention

SUMMARY:
In this study, the researchers will evaluate the efficacy of an intervention using the SALT CONTROL H instrument (an innovative equipment to monitor and control salt) in workers at the University of Porto to reduce dietary salt intake. This is a randomized clinical trial with intervention conducted according to good clinical practice guidelines.

The researchers will randomize 260 workers who meet the eligibility criteria and are enrolled in occupational health appointments. Prior to the intervention, the informed consent of the participants will be obtained and those who agree to participate will be allocated randomly in one of the two arms of the study (control or intervention), with balance of baseline characteristics (sex and hypertension).

The intervention will last for 8 weeks, an individual session of presentation of SALT CONTROL H will be carried out, with explanation of how the equipment works in the culinary preparation with an adequate salt content, will be used an illustrative video and recipes with an adequate salt content; use of SALT CONTROL H at home by the participant to control the use of salt during the cooking process; supervision and enhancement of the use of equipment; daily occurrence log; and the application of a satisfaction questionnaire on the use of SALT CONTROL H. A leaflet will also be delivered about "The new Food Wheel, a guide to the daily food choice!".

Control Group: No intervention will be carried out except the provision of a leaflet on "The new Food Wheel, a guide to the daily food choice!" to the participants.

Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention analysis will cover the following domains: urinary sodium excretion corresponding to a 24 hour urine collection as a proxy for salt intake; 24-hour urinary potassium excretion, sodium:potassium ratio, systolic and diastolic blood pressure, and anthropometric measurements. Urine samples will be collected according to standardized procedures and analyzed by a certified laboratory. Secondary data such as satisfaction questionnaire, daily use of equipment, iodine analysis of salt used and excreted in urine 24h, hydration status, analysis of quality of life and quality of diet will also be analyzed, as well as intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Adults (> 18 years)
* Eat frequently cooked meals at home (> 4 days a week, of which at least 3 Sundays / month)
* Have an occupational health appoitments at São João Hospital
* Reported motivation to control salt consumption

Exclusion Criteria:

* Pregnant
* Subjects with kidney disease,
* Subjects with active infection with an impact on renal function,
* Subjects with urinary incontinence,
* Subjects with acute coronary syndrome,
* Subjects with severe liver disease;
* Subjects with heart failure;
* Subjects who do not use salt for cooking;
* Subjects with hypotension;
* Subjects that work at Faculty that are the Sponsor of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline 24h urinary sodium excretion at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Sodium excretion as a proxy of dietary salt intake

SECONDARY OUTCOMES:
Change from Baseline 24h urinary potassium excretion at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Urinary potassium excretion as a proxy of dietary potassium intake
Change from Baseline Systolic Blood Pressure at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Systolic blood pressure
Change from Baseline Diastolic Blood Pressure at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Diastolic blood pressure
Change from Baseline Hydration Status at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  urinary osmolality (mOsm/kg)
Change from Baseline Perception of quality of life at during and after intervention | Baseline, at 8th intervention week, and 6 months after intervention
  Questionnaire WHOQOL-BREF, results from 0 to 100, higher values represent better perception of quality of life
Change from Baseline Culinary competences at during and after intervention | Baseline, at 8th intervention week, and 6 months after intervention
  Questionnaire, questions scales from 1 to 6 according to culinary competences, higher values represent better culinary competences
Change from Baseline Intestinal Microbiota at after intervention | Baseline and at 8th intervention week
  OTU (operational taxonomy unit) analysis (%)
Change from Baseline Diet Quality at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  HDI (Healthy Diet Indicator), HDI-2015 was calculated as the sum of 7 components (range 0-7) and was classified as follows: high adherence (met 6-7 components), moderate adherence (met 4-5 components), and low adherence (met 0-3 components)
Change from Baseline Knowledges, attitudes and behaviours about salt at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Questionnaire on Knowledge, Attitudes, Behavior toward Dietary Salt and Health from PAHO (n and %)
Change from Baseline Weight at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Weight in kilograms
Change from Baseline Height at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Height in meters
Change from Baseline Fat Mass and Fat Free Mass at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Fat mass (in kg), Fat free mass (in kg)
Change from Baseline Extra and intra cellular water at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Extra and intra cellular water, basal metabolic rate
Change from Baseline Extra and intra cellular water at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Extra and intra cellular water (in kg)
Change from Baseline Basal Metabolic Rate at during and after intervention | Baseline, at the 4th and 8th intervention weeks, and 6 months after intervention
  Basal metabolic rate (in kcal)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Gonçalves, PhD, Principal Investigator — Researcher
Locations (1):
- Carla Gonçalves, Porto, Portugal

IPD SHARING:
Plan to Share IPD: Undecided
In order to promote the quality of the data, they will be introduced by an researcher with delegation of competences by the PI, a verification of double data entry and verification of outliers will be performed. The data will be used for publication of the results by the researchers of the project and for the accomplishment of master's and doctoral thesis.

REFERENCES:
- [Background] Goncalves C, Abreu S, Padrao P, Pinho O, Graca P, Breda J, Santos R, Moreira P. Sodium and potassium urinary excretion and dietary intake: a cross-sectional analysis in adolescents. Food Nutr Res. 2016 Apr 11;60:29442. doi: 10.3402/fnr.v60.29442. eCollection 2016. PMID 27072344
- [Background] Goncalves C, Monteiro S, Padrao P, Rocha A, Abreu S, Pinho O, Moreira P. Salt reduction in vegetable soup does not affect saltiness intensity and liking in the elderly and children. Food Nutr Res. 2014 Oct 6;58. doi: 10.3402/fnr.v58.24825. eCollection 2014. PMID 25317121
- [Background] Moreira P, Sousa AS, Guerra RS, Santos A, Borges N, Afonso C, Amaral TF, Padrao P. Sodium and potassium urinary excretion and their ratio in the elderly: results from the Nutrition UP 65 study. Food Nutr Res. 2018 Feb 27;62. doi: 10.29219/fnr.v62.1288. eCollection 2018. PMID 29545733
- [Derived] Goncalves C, Silva-Santos T, Abreu S, Padrao P, Graca P, Oliveira L, Esteves S, Norton P, Moreira P, Pinho O. Innovative equipment to monitor and control salt usage when cooking at home: iMC SALT research protocol for a randomised controlled trial. BMJ Open. 2020 May 17;10(5):e035898. doi: 10.1136/bmjopen-2019-035898. PMID 32423935